CLINICAL TRIAL: NCT07366203
Title: Clinical Investigation to Evaluate the Use of Adjustable Carbon Fiber Sternal Plates for Sternotomy Closure
Brief Title: Adjustable Carbon Fiber Sternal Plates for Sternotomy Closure
Acronym: FIX IT ALL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NEOS Surgery (Industry)
Collaborators: Fundacio Privada Mon Clinic Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NEO-SC3-2025-01
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Sternotomy Closure,Open Heart Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SC03 plates (Experimental): Adjustable carbon fiber sternal plates
  Interventions: Device: SC03 Plating system
- Wires (Active Comparator): Stainless steel sternal wires
  Interventions: Device: Stainless steel wires

INTERVENTIONS:
Device: SC03 Plating system — Adjustable carbon fiber sternal plates
  Arms: SC03 plates
Device: Stainless steel wires — Nonabsorbable, sterile, surgical sutures used in sternal closure
  Arms: Wires

SUMMARY:
The goal of this clinical trial is to learn if a new medical device (SC03 plates) to close the sternum after a sternotomy in patients that have been operated of a cardiac surgery, is safe and effective. The main question it aims to answer is:

Do patients that have the sternum closed with the SC03 plates present a stable sternum one month after surgery?

Researchers will compare the SC03 plates with stainless steel wires (current standard of care to close the sternum).

Participants will:

* be implanted with the SC03 or stainless steel wires.
* visit the clinic one month and six months after surgery
* Keep a diary of their symptoms and analgesia use

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old.
* Patient who must undergo surgery in which a median or an upper partial sternotomy is indicated.
* Patients capable of giving their voluntary informed consent to participate in the clinical investigation and from whom written consent has been obtained.
* Patient able and willing to meet the protocol requirements and to follow postoperative care instructions

Exclusion Criteria:

* Patient with sternal anomalies, such as bone tumours located in the sternum.
* Patient with limited sternum bone blood supply.
* Patient with suspected or known allergies or intolerances to the implants materials: PEEK, carbon fibre, titanium, stainless steel.
* Patient with severe osteoporosis or other degenerative bone diseases that affect the sternum.
* Pregnant or breastfeeding patient or patient planning to become pregnant during the first 6 months after surgery.
* Patient who is currently using opioid analgesics (e.g., morphine, oxycodone, hydrocodone, fentanyl, tramadol) for the management of chronic or acute pain.
* Patient with diagnosis of dementia with a mental status score (MMSE) < 20.
* Patient with life expectancy lower than 6 months.
* Patient with any other medical process that may compromise or limit the adequate functionality of the implants.
* Patient involved in other interventionist clinical trial or that have been involved in other interventionist clinical trial during the previous 4 weeks.
* Patient with signs of latent or active infection or inflammation on the surgical site.
* Patient with insufficient quantity or quality of sternum bone, or other severe structural bone damage.
* Patient for whom the closure technique cannot ensure sufficient sternal fixation.
* Parasternal sternotomy.
* Patient with intraoperative conditions that may compromise or limit the adequate functionality of the implants or that may prevent the surgeon to use the sternal closure system or that cannot be closed following the product instructions for use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Sternal stability | 1 month post operatively
  Sternal stability measured by clinical assessment using the sternal instability scale (SIS), with grades 0 to 3 where 0 is "Clinically stable sternum" and 3 is "Completely separated sternum - entire length"

SECONDARY OUTCOMES:
Safety of the SC03 Plating System | Perioperative, 1 month and 6 months postoperatively.
  Incidence of Device Deficiencies, AE and SAE with a possible, probable or causal relationship with the device or the procedure.
Reinterventions | 1 month and 6 months postoperatively
  Incidence and cause of surgical reinterventions
Infections | First month and six months postoperatively.
  Incidence of sternal superficial and deep wound infections (mediastinitis)
Sternal dehiscence | First month and six months postoperatively
  Incidence of sternal dehiscence (without infection)
Sternotomy closure duration | Surgery
  Duration of sternotomy closure procedure (minutes)
Easiness of use of the closure method | Surgery
  Surgeon-reported ease of use and satisfaction score (Likert Scale, from 1 to 5)
Sternal Pain | Baseline, 7 days, 1 month and 6 months postoperatively.
  Patient-reported sternal pain at rest and during forced cough, measured by Numerical Rating Scale (0-10)
Analgesia required | Day 7, 1 month and 6 months postoperatively
  Type and cumulative dose of analgesia (total morphine milligram equivalents (MME))
Post-surgery blood loss | 12 hours postoperatively
  Chest tube drainage (mL)
Blood loss | 48 hours after surgery
  Haemoglobin drop (g/dL)
Blood loss | 48 hour after surgery
  Number of administered perioperative blood transfusions of packed red blood cells
Intensive Care Unit stay duration | from surgery date to Intensive care unit discharge date (up to 150 days)]
  Intensive Care Unit stay duration (hours)
hospitalization duration | from surgery date to hospital discharge date (up to 150 days)
  hospitalization duration (days)
sternal stability | 7 days and 6 months postoperatively
  Sternal stability clinically assessed with the sternal instability scale (from 0 to 3)
Upper Limb functional index | Before surgery, one month and 6 months postoperatively
  Patients will assess their upper limbs functional capacity using the Upper Limb functional index (ULFI-Sp)
Quality of life - EQ5D5L | Before surgery, one month and 6 months postoperatively
  Patients will complete the EQ-5D-5L questionnaire
Chest bulging | 1 month after surgery
  Presence of visible bulging related to the sternal closure method on the sternotomy area
Pulmonary function | Baseline, day 7 and 1 month postoperatively
  Pulmonary function (FVC, FEV1 and FEV1/FVC) measured by spirometry

IPD SHARING:
Plan to Share IPD: No